CLINICAL TRIAL: NCT04937036
Title: Evaluation of Impact of Bruxism Related Arousals on Cardiovascular Risk in Co-morbid Insomnia and Sleep Apnea (COMISA)
Brief Title: Impact of Bruxism Related Arousals on Cardiovascular Risk in Co-morbid Insomnia and Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Smardz, Investigator, Wroclaw Medical University
Other Study IDs: WMU1/2021
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Sleep Apnea; Sleep Bruxism; Sleep Disorder; Insomnia; Comorbidities and Coexisting Conditions; Cardiovascular Diseases
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Bruxism; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Cardiovascular Diseases | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COMISA group: Patients with diagnosed COMISA.
  Interventions: Diagnostic Test: Polysomnography
- Healthy controlls: Healthy indyviduals.
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Each of the patients will undergo polysomnography

SUMMARY:
Sleep disordered breathing is a common and serious health problem. According to epidemiological data, it may affect about 20% of adult population. The majority is not aware of the disease. The most common sleep disorder is obstructive sleep apnea (OSA). The essence of OSA are the episodes of airway obstruction repeated many times during sleep, as a result of which the level of partial oxygen in the blood decreases. Apnea episodes end up waking from sleep, causing sleep fragmentation, deep sleep and REM deficiency. Frequent complications of OSA are hypertension, stroke, cardiac arrhythmia, coronary artery disease and pulmonary hypertension.

Comorbid Insomnia and Sleep Apnea (COMISA) is a highly prevalent and debilitating disorder that causes additional disturbances in sleep, daytime functioning, and quality of life for patients, and is a significant diagnostic and therapeutic problem for clinicians. Although the presence of COMISA was first noticed by Christian Guilleminault and his colleagues in 1973, it received very little research attention for almost three decades. There is still lack ofclinical trials concerning this topic.

An additional problem in apnea patients is the increased incidence of bruxism. Bruxism is associated with increased masticatory muscle activity during sleep, which may be phased or tonic. It is estimated that the incidence of bruxism in the adult population is 13%. The most common symptoms of bruxism include: pathological wear and tooth sensitivity, damage to the periodontium and oral mucosa, muscle pain in the stomatognathic system, headaches and damage to prosthetic restorations. However, the symptoms of bruxism can go unnoticed for a long time, leaving patients often unaware of the problem.

The aim of this project is:

1. to determine the prevalence of sleep bruxism in COMISA, OSA and insomnia,
2. to examine of arousals (type, frequency) in COMISA, OSA and insomnia,
3. to investigate the relationship between arousals and blood pressure values and variability, arrhythmias, sinus rhythm variability, vascular endothelial dysfunction, cardiovascular risk in COMISA, OSA and insomnia.

DETAILED DESCRIPTION:
I. Introduction

Sleep disordered breathing is a common and serious health problem. According to epidemiological data, it may affect about 20% of the adult population, the majority is not aware of the disease. The most common sleep disorder is obstructive sleep apnea (OSA). The essence of OSA are the episodes of airway obstruction repeated many times during sleep, as a result of which the level of partial oxygen in the blood decreases. Apnea episodes end up with arousal, causing sleep fragmentation, deep sleep and REM deficiency. The consequence of episodes of OSA and fragmentation of sleep is ineffective, non-restful sleep, pathological daytime sleepiness, shortness of breath or choking. Fragmentation of sleep and repeated episodes of hypoxia result in a deterioration of the quality of life, chronic fatigue, and an increased risk of road accidents. The immediate consequences of apnea are hypoxia, awakening, increased heart rate, and an increase in blood pressure. Common complications of OSA include high blood pressure, stroke, arrhythmias, coronary artery disease, pulmonary hypertension, and heart failure. Untreated OSA increases the risk of premature death, especially in men under 50, contributing to the development of vascular endothelial dysfunction and increasing cardiovascular risk.

Comorbid Insomnia and Sleep Apnea (COMISA) is a highly prevalent and debilitating disorder that causes additional disturbances in sleep, daytime functioning, and quality of life for patients, and is a significant diagnostic and therapeutic problem for clinicians. Although the presence of COMISA was first noticed by Christian Guilleminault and his colleagues in 1973, it received very little research attention for almost three decades. There is still lack ofclinical trials concerning this topic.

An additional problem in OSA patients is the increased incidence of bruxism. Bruxism is associated with increased masticatory muscle activity during sleep, which may be phasic or tonic. It is estimated that the incidence of bruxism in the adult population is 13%. The most common symptoms of bruxism include: pathological wear and tooth sensitivity, damage to the periodontium and oral mucosa, muscle pain, headaches and damage to prosthetic restorations. However, the symptoms of bruxism can go unnoticed for a long time, leaving patients often unaware of the problem. There are two different types of bruxism: sleep bruxism (SB) and awake bruxism (AB). The etiology of bruxism is multifactorial and not fully understood, it is believed that it may be modulated by biological, psychological and exogenous factors. Bruxism may also be a protective factor in patients with disordered breathing during sleep. A key aspect of this relationship is likely related to arousals.

So far, it has not been possible to clearly define the exact cause-and-effect relationship between obstructive sleep apnea, insomnia and sleep bruxism. The relationship with cardiovascular risk is also unclear.More research is needed to clarify the relationship between these phenomena.

II. Aim

The aim of this project is:

1. to determine the prevalence of sleep bruxism in COMISA, OSA and insomnia,
2. to examine of arousals (type, frequency) in COMISA, OSA and insomnia,
3. to investigate the relationship between arousals and blood pressure values and variability, arrhythmias, sinus rhythm variability, vascular endothelial dysfunction, cardiovascular risk in COMISA, OSA and insomnia.

III. Methods

The project will take place at the Sleep Laboratory at the Department and Clinic of Internal Medicine, Occupational Diseases, Hypertension and Clinical Oncology of the Wroclaw Medical University. About 120 patients will be examined, referred to the Department and Clinic of Internal Medicine, Occupational Diseases, Hypertension and Clinical Oncology due to suspected COMISA and sleep apnea.

Polysomnograms will be assessed in 30 second epochs, according to standard sleep criteria. The PSG results will include data on sleep latency, total sleep time (TST), and sleep efficiency (%), as well as an assessment of N1, N2, N3, and REM sleep stages. Pathological respiratory events will be assessed according to the American Academy of Sleep Medicine standards. An apnea will be defined as the lack of airflow through the airways for more than 10 seconds. Hypopnea will be defined as a reduction in respiratory amplitude by more than 30% for more than 10 seconds, followed by blood desaturation by more than 3% or subsequent arousal. Also, limb movements and types of arousals (including spontaneous and related to limb movements, periodic limb movements, respiratory events and bruxism) and RERA will be assessed. The activity of the masticatory muscles will be assessed on the basis of the EMG recording from the electrodes placed in the area of masseter muscles. Bruxism will be assessed both quantitatively and qualitatively.

In each patient, diagnostics will also be extended to ambulatory blood pressure measurement (ABPM), central blood pressure measurement and EKG Holter. Each patient will give the blood sample to measure inflammatory markers (interleukin, TNF alpha, fibrinogen, CRP), lipid profile (TGL, cholesterol, LDL, HDL), creatinine, glucose, blood count, electrolytes and markers of vascular endothelial dysfunction in serum. Each patient will have their cardiovascular risk assessed (SCORE). Patients will also fill in the questionnaires: Epworth Sleepiness Scale, STOP-bang questionnaire, author's questionnaire on cardiovascular risk factors, Pittsburg Sleep Quality Index, Munich Chronotype Questionnaire, Insomnia Severity Index, Graded Chronic Pain Scale , Patient Health Questionnaire - 9, Perceived Stress Scale - 10, Generalized Anxiety Disorder - 7 questionnaire, the Athens Insomnia Scale, Satisfaction With Life Scale, Somatic Symptom Scale - 8, Central Sensitization Inventory and Migraine Disability Assessment Test (MIDAS).

IV. Expected effects

Participation in the project will enable patients with COMISA syndrome detailed sleep diagnostics, which is extremely beneficial due to the fact that access to polysomnographic assessment is quite limited. In addition, the research will allow to determine the potential cause-and-effect relationship between bruxism and cardiovascular risk in patients with COMISA syndrome, which in the future will contribute to more effective diagnostics and therapy of all described entities.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years old
* suspicion of COMISA

Exclusion Criteria:

* age under 18
* age over 75
* terminal general diseases
* severe mental disorders
* taking drugs that could falsify polysomnography
* confirmed alcoholism
* drug addiction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of COMISA referred to the Department of Internal Medicine, Occupational Diseases, Hypertension and Clinical Oncology operating at the Wroclaw Medical University. Healthy controls.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
The incidence of sleep bruxism in obstructive sleep apnea, insomnia and COMISA. | 01.07.2021-31.12.2022
  Each participant will undergo audio-video polysomnography to assess sleep bruxism, sleep-related breathing disorders and other sleep parameters. Polysomnograms will be evaluated in a 30-second contributions, according to standard sleep criteria.
The meaning of arousals in relationships between sleep bruxism, obstructive sleep apnea, insomnia and COMISA, | 01.07.2021-31.12.2022
  Each participant will undergo audio-video polysomnography to assess sleep bruxism, sleep-related breathing disorders and other sleep parameters (especially arousals: type, frequency).

SECONDARY OUTCOMES:
Relationship between sleep bruxism, obstructive sleep apnea and insomnia assessed by Athens Insomnia Scale. | 01.07.2021-31.12.2022
  Each participant will fill in Athens Insomnia Scale (AIS). Each item is rated on a 4-point numerical rating scale (NRS; where 0= no problem at all and 3= very serious problem). Total scores range from 0 to 24 in the AIS-8. Higher scores in these AIS measures indicate that responders have severe insomnia symptoms.
Relationship between sleep bruxism, obstructive sleep apnea and insomnia assessed by Insomnia Severity Index. | 01.07.2021-31.12.2022
  Each participant will fill in Insomnia Severity Scale. Questionnaire contains 5 questions, scored from 0 to 4 depending on the severity of ailments. Minimal score is 0, maximal score is 20. A total point value of up to 10 is considered the norm, while a score above 14 points indicates clinically significant insomnia.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and pain assessed by Graded Chronic Pain Scale. | 01.07.2021-31.12.2022
  Each participant will fill in Graded Chronic Pain Scale. Scoring Criteria for Grading Chronic Pain Severity: Characteristic Pain Intensity is a 0 to 100 score derived from Questions 1 through 3:Mean (Pain Right Now, Worst Pain, Average Pain) X 10. Disability Score is 0 to 100score derived from Questions 4 through 6:Mean (Daily Activities, Social Activities, Work Activities) X 10. Disability Points: Add the indicated points for Disability Days (Question 7)and for Disability Score. Classification: GRADE 0- No TMD pain in prior 6 months. GRADE I-Low Intensity Characteristic Pain Intensity<50, Low Disability<3 Disability Point. GRADE II -High Intensity Characteristic Pain Intensity >50, LowDisability<3 Disability Points. GRADE III- High Disability3 to 4 Disability Points, Moderately Limiting (Regardless of Characteristic Pain Intensity). GRADE IV- High Disability 5 to 6 Disability Points, Severely Limiting (Regardless of Characteristic Pain Intensity).
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and depression assessed by Patient Health Questionnaire - 9. | 01.07.2021-31.12.2022
  Each participant will fill in Patient Health Questionnaire - 9. PHQ-9 total score for the nine items ranges from 0 to 27.Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and sleep quality assessed by Pittsburgh Sleep Quality Index - a self-report questionnaire that assesses sleep quality over a 1-month time interval. | 01.07.2021-31.12.2022
  Each participant will fill in Patient Health Questionnaire - 9. PHQ-9 total score for the nine items ranges from 0 to 27.Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Relationship between sleep bruxism, insomnia and apnea risk assessed by STOP-Bang. | 01.07.2021-31.12.2022
  Each participant will fill in STOP-Bang questionnaire. The total score ranges from 0 to 8. The lower the score is, the lower the risk of occurrence Obstructive Sleep Apnea (OSA).
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and perceived stress assessed by Perceived Stress Scale - 10. | 01.07.2021-31.12.2022
  Each participant will fill in Perceived Stress Scale -10. Scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items. It can range from 0 to 40. Scores ranging from 0-13 would be considered low stress,14-26 would be considered moderate stress, 27-40 would be considered high perceived stress.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and anxiety assessed by Generalized Anxiety Disorder -7. | 01.07.2021-31.12.2022
  Each participant will fill in Generalized Anxiety Disorder -7 that consists of 7 items. Total score ranges 0-21 points. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and quality of sleep assessed by Epworth Sleepiness Scale. | 01.07.2021-31.12.2022
  Each participant will fill in Epworth Sleepiness Scale. The questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 to 3 for eight different situations that most people engage in during their daily lives, though not necessarily every day. The scores for the eight questions are added together to obtain a single number. A number in the 0-9 range is considered to be normal while a number in the 10-24 range indicates that expert medical advice should be sought. For instance, scores of 11-15 are shown to indicate the possibility of mild to moderate sleep apnea, where a score of 16 and above indicates the possibility of severe sleep apnea or narcolepsy.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and satisfaction with life assessed by Satisfaction With Life Scale. | 01.07.2021-31.12.2022
  Each participant will fill in Satisfaction With Life Scale (SWLS). The SWLS is a 7-point Likert style response scale. The possible range of scores is 5-35, with a score of 20 representing a neutral point on the scale. Scores between 5-9 indicate the respondent is extremely dissatisfied with life, whereas scores between 31-35 indicate the respondent is extremely satisfied.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and somatic symptoms assessed by Somatic Symptom Scale - 8. | 01.07.2021-31.12.2022
  Each participant will fill in the Somatic Symptom Scale - 8 (SSS-8) which is a brief self-report questionnaire used to assess somatic symptom burden. It measures the perceived burden of common somatic symptoms. These symptoms were originally chosen to reflect common symptoms in primary care but they are relevant for a large number of diseases and mental disorders. Scoring: 0-3: no to minimal, 4-7: low, 8-11: medium,12-15: high,16-32: very high.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and central sensitization assessed by Central Sensitization Inventory. | 01.07.2021-31.12.2022
  Each participant will fill in the Central Sensitisation Inventory (CSI) which is a self-report outcome measure designed to identify patients who have symptoms that may be related to central sensitisation or central sensitivity syndromes. Part A includes 25 questions related to common CSS symptoms. Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and chronotype assessed by Munich Chronotype Questionnaire (MCTQ). | 01.07.2021-31.12.2022
  Each participant will fill in Munich Chronotype Questionnaire (MCTQ). Questions about work day and free day sleep schedules, work details, and lifestyle provide data to aid in the understanding of how biological clocks work in social life, such as Roenneberg's conclusions of social jetlag. The MCTQ categorizes each participant into one of seven chronotype groups, and utilizes data on participants' midsleep phase and sleep debt to survey what "type" of sleeper each person is. From these data, the MCTQ offers methods to make up for sleep debt (if any), and offers suggestions on what to do to wake up earlier or sleep later
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and headache assessed by Migraine Disability Assessment Test (MIDAS). | 01.07.2021-31.12.2022
  The Migraine Disability Assessment Test (MIDAS) is a test used by doctors to determine how severely migraines affect a patient's life. Patients are asked questions about the frequency and duration of their headaches, as well as how often these headaches limited their ability to participate in activities at work, at school, or at home.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and cardiovascular risk assessed by ambulatory blood pressure measurement (ABPM). | 01.07.2021-31.12.2022
  Cardiovascular risk will be assessed in each participant using ambulatory blood pressure measurement (ABPM).
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and cardiovascular risk assessed by ECG Holter. | 01.07.2021-31.12.2022
  Cardiovascular risk will be assessed in each participant using ECG Holter.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and cardiovascular risk assessed by central blood pressure measurement. | 01.07.2021-31.12.2022
  Cardiovascular risk will be assessed in each participant using central blood pressure measurement.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and cardiovascular risk assessed by cardiovascular risk assessment tool (SCORE). | 01.07.2021-31.12.2022
  Cardiovascular risk will be assessed in each participant using SCORE.
Relationship between sleep bruxism, obstructive sleep apnea, COMISA and blood parameters assessed by blood tests. | 01.07.2021-31.12.2022
  Each participant will undergo blood tests to assess: inflammatory markers (interleukin, TNF alpha, fibrinogen, CRP), lipid profile (TGL, cholesterol, LDL, HDL), creatinine, glucose, blood count, electrolytes and markers of vascular endothelial dysfunction in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Martynowicz, Associate professor, Principal Investigator — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided